CLINICAL TRIAL: NCT06529419
Title: A Phase 2b, Randomised, Double-Blind, Placebo-Controlled Dose Range-Finding Study to Assess Efficacy and Safety of Multiple Dose Levels of Inhaled AZD8630 Given Once Daily for 12 Weeks in Adults With Uncontrolled Asthma at Risk of Exacerbations (LEVANTE)
Brief Title: A Dose Range-Finding Study to Assess the Efficacy and Safety of Multiple Dose Levels of AZD8630 in Adults With Uncontrolled Asthma at Risk of Exacerbations
Acronym: Levante
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6830C00003
Record Dates: First submitted 2024-07-15; First posted 2024-07-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: This is a parallel-group treatment study with 4 arms that is patient and Investigator blinded. Patients will be randomly assigned in a 1:1:1:1 ratio to one of the 4 treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- AZD8630 dose A (Experimental): Inhaled AZD8630 administered at a dose A
  Interventions: Drug: AZD8630; Device: Inhaler
- AZD8630 dose B (Experimental): Inhaled AZD8630 administered at a dose B
  Interventions: Drug: AZD8630; Device: Inhaler
- AZD8630 dose C (Experimental): Inhaled AZD8630 administered at a dose C
  Interventions: Drug: AZD8630; Device: Inhaler
- Placebo (Placebo Comparator): Inhaled placebo
  Interventions: Drug: Placebo; Device: Inhaler

INTERVENTIONS:
Drug: AZD8630 — The drug will be administered by inhalation
  Arms: AZD8630 dose A; AZD8630 dose B; AZD8630 dose C
Drug: Placebo — The placebo will be administered by inhalation
  Arms: Placebo
Device: Inhaler — The drug/placebo will be administered by inhalation using the inhaler

SUMMARY:
A dose range-finding study to assess the efficacy and safety of multiple dose levels of AZD8630 administered via a dry powder inhaler in adults with uncontrolled asthma at risk of exacerbations, receiving medium -to -high dose inhaled corticosteroid (ICS)/long-acting β2-agonist (LABA).

DETAILED DESCRIPTION:
This is a Phase II, randomised, placebo-controlled, double-blind, dose range-finding, multi-centre study to assess the efficacy and safety of inhaled AZD8630 administered at 3 doses via an inhaler in adult patients with uncontrolled asthma, at risk of an exacerbation. The study duration up to 57 weeks for participants in the optional safety extension study and up to 17 weeks for those not included. The maximal treatment period is up to 52 weeks.

This study will be conducted in approximately 220 centres in 20-25 countries. Approximately 516 patients will be randomised globally

ELIGIBILITY:
Principal inclusion criteria (abbreviated):

1. Patient must be 18 to 80 years of age inclusive
2. Documented physician diagnosis of asthma for at least 12 months, with objective evidence of asthma (spirometric, bronchial challenge, exercise challenge or therapeutic response) within the last 5 years

4. Uncontrolled asthma (i.e. ACQ-6 ≥ 1.5)

5. Pre-BD FEV1 ≥ 40%

7. A history of asthma exacerbations within the last 12 months

8. & 9. Compliant with asthma background mediation, daily ePROs and daily home spirometry.

10. BMI within the range 18-37 kg/m2 (inclusive)

11. Female patients of child bearing potential must not be pregnant and agree to use highly effective contraception.

12. Male patients and their female partners of childbearing potential must agree to use highly effective contraception.

13. Capable of giving signed informed consent.

Principal exclusion criteria (abbreviated):

1. History of life-threatening asthma
2. Recently completed treatment for respiratory infection and/or asthma exacerbation
3. Clinically important pulmonary disease other than asthma; including but not limited to those with co-existent chronic obstructive pulmonary disease.
4. Any disorder that is not stable in the opinion of the Investigator and could:

   1. Affect the safety of the patient throughout the study
   2. Influence the findings of the study or their interpretation
   3. Impede the patient's ability to complete the entire duration of study
5. Patients who, in the opinion of the Investigator, have evidence of active TB or are currently on treatment for active or latent TB.
6. Medical history of or treatment for hepatitis B or hepatitis C, except for cured hepatitis C
7. Patients with history of HIV infection or who test positive for HIV.
8. Congenital long QT syndrome or prolonged QTcF > 470 ms or history of QT prolongation associated with other medications that required discontinuation of that medication.
9. Current untreated or uncontrolled arrhythmia.
10. Patients with recent myocardial infarction, unstable angina pectoris, stroke, percutaneous coronary intervention or coronary artery bypass grafting.
11. A helminth parasitic infection diagnosed that has not been treated, or has not responded to SoC therapy.
12. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months ago.
13. Known history of drug or alcohol abuse within 12 months, that in the Investigator's opinion would preclude participation in the study.
14. Current diagnosis of cancer or unresectable cancer that has not been in complete remission for at least 5 years.
15. Any other clinically relevant abnormal findings that in the opinion of the Investigator or medical monitor might compromise the safety of the patient in the study or interfere with evaluation of the study intervention.
16. Treatment with marketed or investigational biologics within 4 months or a minimum of 5 half-lives.
17. Treatment with Systemic steroids within 4 weeks.
18. Chronic oral or systemic CS use for asthma or for any other indication (with the exception of stable replacement therapy in adrenal insufficiency).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Time to first CompEx Asthma event | 12 weeks
  The CompEx Asthma is a composite endpoint for exacerbations that captures asthma-worsening episodes based on combination of diary events (worsening in daily PEF, asthma symptoms and rescue medication use) plus severe asthma exacerbation events. Diary events are defined by threshold and slope criteria using the following morning/evening diary variables:
  * PEF
  * Asthma symptom score (0 to 3)
  * Use of rescue medication

SECONDARY OUTCOMES:
Pre-BD FEV1 | 12 weeks
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second.
ACQ-6: | 12 weeks
  Change from baseline in the Asthma Control Questionnaire 6 (ACQ-6). The ACQ-6 has 6 questions (regarding asthma symptoms and rescue bronchodilator use). Answering the questions results in a score out of 6. A Score of 0 indicates complete control and 6 reflects severely uncontrolled disease
AQLQ12+ | 12 weeks
  Change from baseline in the Asthma Quality of Life Questionnaire for 12 Years and Older. The AQLQ12+ includes 32 questions grouped into four domains: symptoms; activity limitations; emotional function; and, environmental stimuli. Each question is scored on a seven-point Likert scale, which ranges from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean of all questions, and the four domain scores are the means of the scores for the questions in the respective domains
SGRQ | 12 weeks
  Change from baseline in the St. George's Respiratory Questionnaire. The SGRQ includes 50 questions grouped into two parts: Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
FeNO | 12 weeks
  Change from baseline to: FeNO: Weeks 1, 2, 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo, Principal Investigator — Univeristy of Michigan Hospital, Ann Arbor, MI, US
Locations (179):
- United States (44):
  - Research Site, Mesa, Arizona
  - Research Site, Huntington Beach, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Niguel, California
  - Research Site, Lancaster, California
  - Research Site, Long Beach, California
  - Research Site, San Jose, California
  - Research Site, New Haven, Connecticut
  - Research Site, DeBary, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jensen Beach, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lilburn, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Ames, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Methuen, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Riverdale, New Jersey
  - Research Site, Middletown, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Beavercreek, Ohio
  - Research Site, Lima, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Horsham, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, McKinney, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, American Fork, Utah
  - Research Site, Roy, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Hampton, Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (9):
  - Research Site, Alberdi
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Mar del Plata
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Belgium (3):
  - Research Site, Duffel
  - Research Site, Mechelen
  - Research Site, Namur
- Chile (5):
  - Research Site, Chile
  - Research Site, Curicó
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Viña del Mar
- China (19):
  - Research Site, Baotou
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Xuzhou
- Czechia (8):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jindřichův Hradec
  - Research Site, Kralupy nad Vltavou
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Varnsdorf
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense
  - Research Site, Roskilde
  - Research Site, Vejle
- France (5):
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Reims
- Germany (8):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
- Research Site, Hong Kong, Hong Kong
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (3):
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Roma
- Japan (17):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiratsuka-shi
  - Research Site, Hiroshima
  - Research Site, Kitakyushu
  - Research Site, Kusatsu-shi
  - Research Site, Maebashi
  - Research Site, Meguro-ku
  - Research Site, Mizunami-shi
  - Research Site, Nankoku-shi
  - Research Site, Niigata
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Toyoake-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Monterrey
  - Research Site, Villahermosa
- Netherlands (2):
  - Research Site, Alkmaar
  - Research Site, Amersfoort
- Slovakia (6):
  - Research Site, Kežmarok
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Prešov
  - Research Site, Topoľčany
  - Research Site, Žilina
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Observatory
  - Research Site, Somerset West
  - Research Site, Tygervalley
- South Korea (2):
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Santander
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Altındağ-Ankara
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Kırıkkale
  - Research Site, Mersin
- Ukraine (6):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Bradford
  - Research Site, Liverpool
  - Research Site, Portsmouth